CLINICAL TRIAL: NCT04841096
Title: Efficacy and Safety of the Oral Combined Therapy Glimepiride / Vildagliptin / Metformin in Patients With Type 2 Diabetes With Dual Treatment Failure
Brief Title: Oral Combination of Glimepiride/Vildagliptin/Metformin in Patients With T2D and Dual Treatment Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SIL-30013-III-20(1)
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes; Combine therapy; Hypoglycemic agents
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A1: Glimepiride (1mg) / Vildagliptin (50mg) / Metformin (500mg). (Experimental): Tablets, orally, once a day. Initial dose for the first 45 days of intervention.
  Interventions: Drug: A1=Glimepiride / Vildagliptin / Metformin (1 mg/ 50 mg/ 500 mg)
- Group B1: Glimepiride (1mg) / Vildagliptin (50mg) / Metformin (500mg) (Experimental): Tablets, orally, once a day. Initial dose for the first 45 days of intervention.
  Interventions: Drug: B2=Glimepiride / Vildagliptin / Metformin (1 mg/ 50 mg/ 500 mg)
- Group A2: Glimepiride (2mg) / Vildagliptin (50mg) / Metformin (1000mg) (Experimental): Tablets, orally, once a day. Dose escalation if the patients meets established criteria.
  Interventions: Drug: (A2) Glimepiride/Vildagliptin/Metformin
- Group B2: Glimepiride (4mg) / Vildagliptin (50mg) / Metformin (1000mg) (Experimental): Tablets, orally, once a day. Dose escalation if the patients meets established criteria.
  Interventions: Drug: (B2) Glimepiride/Vildagliptin/Metformin

INTERVENTIONS:
Drug: A1=Glimepiride / Vildagliptin / Metformin (1 mg/ 50 mg/ 500 mg) — Take one tablet of the prescribed dose of the investigational drug by mouth, preferably with food and in the morning. Initial dose for the first 45 days of intervention.
  Other Names: (A1) Glimepiride/Vildagliptin/Metformin
  Arms: Group A1: Glimepiride (1mg) / Vildagliptin (50mg) / Metformin (500mg).
Drug: B2=Glimepiride / Vildagliptin / Metformin (1 mg/ 50 mg/ 500 mg) — take one tablet of the prescribed dose of the investigational drug by mouth, preferably with food and in the morning. Initial dose for the first 45 days of intervention.
  Other Names: (B1) Glimepiride/Vildagliptin/Metformin
  Arms: Group B1: Glimepiride (1mg) / Vildagliptin (50mg) / Metformin (500mg)
Drug: (A2) Glimepiride/Vildagliptin/Metformin — Take one tablet of the prescribed dose of the investigational drug by mouth, preferably with food and in the morning. Escalation dose in cause the patient meets established criteria.
  Other Names: A2=Glimepiride / Vildagliptin / Metformin (2 mg/ 50 mg/ 1000 mg)
  Arms: Group A2: Glimepiride (2mg) / Vildagliptin (50mg) / Metformin (1000mg)
Drug: (B2) Glimepiride/Vildagliptin/Metformin — Take one tablet of the prescribed dose of the investigational drug by mouth, preferably with food and in the morning. Escalation dose in cause the patient meets established criteria.
  Other Names: B2=Glimepiride / Vildagliptin / Metformin (4 mg/ 50 mg/ 1000 mg)
  Arms: Group B2: Glimepiride (4mg) / Vildagliptin (50mg) / Metformin (1000mg)

SUMMARY:
Phase IIIb, randomized, multicenter, double-blind, prospective study to evaluate the efficacy and safety of a daily fixed-dose combination of glimepiride / vildagliptin / metformin in patients with type 2 diabetes with a history of dual treatment failure and combined or individual oral antidiabetics with SGLT2 / Metformin, Biguanide / Sulfonylurea, Sulfonylurea / iDPP4 or Biguanide / iDPP4. To evaluate the changes in the percentage of HbA1c at 3 and 6 months with regard to their baseline measurement.

DETAILED DESCRIPTION:
To achieve glycemic control goals, a combination of medications with complementary mechanisms of action, with fasting and postprandial effects, may be required to achieve and maintain clinically acceptable glycemic control in some patients. A fixed combination of two or more therapeutic agents with complementary mechanisms of action makes it possible to optimize compliance and adherence to treatment among patients with T2D because it is administered once a day with the same efficacy of the separate components, but with fewer gastrointestinal effects. This is reflected in a reduction in HA1c and a lower evolution to long-term complications of T2D. Phase IIIb, randomized, multicenter, double-blind, prospective study to evaluate the efficacy and safety of a daily fixed-dose combination of glimepiride / vildagliptin / metformin in patients with type 2 diabetes with a history of dual treatment failure and combined or individual oral antidiabetics with SGLT2 / Metformin, Biguanide / Sulfonylurea, Sulfonylurea / iDPP4 or Biguanide / iDPP4.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female.
* Age >18 years old at the beginning of the study.
* Diagnosis of type 2 diabetes prior to the start of the study.
* Therapeutic failure to a dual treatment with SGLT2 / Metformin, Biguanide / Sulfonylurea, Sulfonylurea / iDPP4, Biguanide / iDPP4.
* HbA1c ≥ 7.5% and ≤ 11% during screening tests.
* Women of childbearing potential using a contraceptive method (barrier, oral hormonal, injectable, subdermal) or naturally or surgically sterile in menopause.
* Subject agree to participate in the study and give informed consent in writing.

Exclusion Criteria:

* The drug is contraindicated for medical reasons.
* History of Type 1 Diabetes Mellitus.
* History of metabolic complications such as ketoacidosis or nonketotic hyperosmolar state.
* History of gastric bariatric surgery or gastric band in the last year.
* History of drug or alcohol abuse in the past year.
* Body Mass Index <20 kg/m2 and >40 kg/m2.
* Acute or severe renal dysfunction (glomerular filtration <30 ml / min / 1.72 m2).
* History of chronic liver disease or ALT and / or AST ≥3 times the normal upper limit and / or Total Bilirubin> 2.5 times the upper limit of normal, or GGT ≥3 times the upper limit of normal.
* Pregnant and / or lactating women.
* The patient is participating in another clinical study involving an investigational treatment or participated in one in the previous 4 weeks.
* At medical criteria, a disease that affects the prognosis and prevents outpatient management, for example, but not restricted to: end-stage cancer, kidney, heart, respiratory or liver failure, mental illness, with scheduled surgical or hospital procedures.
* Be a patient with a working relationship with the main researcher or the research center or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Compare changes in HbA1 | baseline, 3 and 6 months of treatment
  Mean change in HbA1c
Proportion of patients who change their HbA1c concentration | baseline, 3 and 6 months of treatment
  Proportion of patients who change their HbA1c by at least 1 percent
Mean difference change between groups in HbA1c concentration | baseline, 3 and 6 months of treatment
  Difference greater than 0.3 between group A and B HbA1c concentration

SECONDARY OUTCOMES:
Mean glucose change | baseline, 3 and 6 months of treatment
  Compare changes in glucose between baseline, 3 and 6 months of treatment
Incidence of adverse events and reactions | baseline, 3 and 6 months of treatment
  Description of al the adverse events and reactions presented during the study

CONTACTS AND LOCATIONS:
Overall Officials: Salvador Pérez Jaime, M.D, Principal Investigator — Centro de Investigación Médica Aguascalientes (Red OSMO); Juan A Becerra Hernández, M.D, Principal Investigator — Centro de Investigación y Avances Médicos Especializados (Red OSMO); Ana L Flores Barranco, M.D, Principal Investigator — Oaxaca Site Management Organization SC. (Red OSMOS); Abraham S Álvarez, M.D, Principal Investigator — Oncológico Potosino (Red OSMO); Victor C Bohórquez López, M.D, Principal Investigator — Mérida Investigación Clínica (Red OSMO)
Locations (5):
- Mexico (5):
  - Centro de Investigación y Avances Médicos Especializados, Cancún, Quintana Roo
  - Mérida Investigación Clínica, Mérida, Yucatán
  - Centro de Investigación Médica Aguascalientes, Aguascalientes
  - Oaxaca Site Management Organization SC., Oaxaca City
  - Oncológico Potosino, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2020. Diabetes Care. 2020 Jan;43(Suppl 1):S14-S31. doi: 10.2337/dc20-S002. PMID 31862745
- [Background] Cahn A, Raz I, Kleinman Y, Balicer R, Hoshen M, Lieberman N, Brenig N, Del Prato S, Cefalu WT. Clinical Assessment of Individualized Glycemic Goals in Patients With Type 2 Diabetes: Formulation of an Algorithm Based on a Survey Among Leading Worldwide Diabetologists. Diabetes Care. 2015 Dec;38(12):2293-300. doi: 10.2337/dc15-0187. Epub 2015 Oct 30. PMID 26519337
- [Background] Cramer JA. A systematic review of adherence with medications for diabetes. Diabetes Care. 2004 May;27(5):1218-24. doi: 10.2337/diacare.27.5.1218. PMID 15111553
- [Background] Rubin RR. Adherence to pharmacologic therapy in patients with type 2 diabetes mellitus. Am J Med. 2005 May;118 Suppl 5A:27S-34S. doi: 10.1016/j.amjmed.2005.04.012. PMID 15850551
- [Background] Khunti K, Kosiborod M, Ray KK. Legacy benefits of blood glucose, blood pressure and lipid control in individuals with diabetes and cardiovascular disease: Time to overcome multifactorial therapeutic inertia? Diabetes Obes Metab. 2018 Jun;20(6):1337-1341. doi: 10.1111/dom.13243. Epub 2018 Mar 11. PMID 29405543
- [Background] Orozco-Beltran D, Mata-Cases M, Artola S, Conthe P, Mediavilla J, Miranda C. [Adherence of Type 2 Diabetes Mellitus approach: Current situation and possible solutions]. Aten Primaria. 2016 Jun-Jul;48(6):406-20. doi: 10.1016/j.aprim.2015.09.001. Epub 2016 Jan 13. Spanish. PMID 26775266
- [Background] Garber AJ, Handelsman Y, Grunberger G, Einhorn D, Abrahamson MJ, Barzilay JI, Blonde L, Bush MA, DeFronzo RA, Garber JR, Garvey WT, Hirsch IB, Jellinger PS, McGill JB, Mechanick JI, Perreault L, Rosenblit PD, Samson S, Umpierrez GE. CONSENSUS STATEMENT BY THE AMERICAN ASSOCIATION OF CLINICAL ENDOCRINOLOGISTS AND AMERICAN COLLEGE OF ENDOCRINOLOGY ON THE COMPREHENSIVE TYPE 2 DIABETES MANAGEMENT ALGORITHM - 2020 EXECUTIVE SUMMARY. Endocr Pract. 2020 Jan;26(1):107-139. doi: 10.4158/CS-2019-0472. No abstract available. PMID 32022600
- [Background] Lukashevich V, Del Prato S, Araga M, Kothny W. Efficacy and safety of vildagliptin in patients with type 2 diabetes mellitus inadequately controlled with dual combination of metformin and sulphonylurea. Diabetes Obes Metab. 2014 May;16(5):403-9. doi: 10.1111/dom.12229. Epub 2013 Dec 2. PMID 24199686
- [Background] Maruthur NM, Tseng E, Hutfless S, Wilson LM, Suarez-Cuervo C, Berger Z, Chu Y, Iyoha E, Segal JB, Bolen S. Diabetes Medications as Monotherapy or Metformin-Based Combination Therapy for Type 2 Diabetes: A Systematic Review and Meta-analysis. Ann Intern Med. 2016 Jun 7;164(11):740-51. doi: 10.7326/M15-2650. Epub 2016 Apr 19. PMID 27088241
- [Background] Dennis JM, Henley WE, Weedon MN, Lonergan M, Rodgers LR, Jones AG, Hamilton WT, Sattar N, Janmohamed S, Holman RR, Pearson ER, Shields BM, Hattersley AT; MASTERMIND Consortium. Sex and BMI Alter the Benefits and Risks of Sulfonylureas and Thiazolidinediones in Type 2 Diabetes: A Framework for Evaluating Stratification Using Routine Clinical and Individual Trial Data. Diabetes Care. 2018 Sep;41(9):1844-1853. doi: 10.2337/dc18-0344. Epub 2018 Aug 2. PMID 30072404
- [Background] Bianchi C, Daniele G, Dardano A, Miccoli R, Del Prato S. Early Combination Therapy with Oral Glucose-Lowering Agents in Type 2 Diabetes. Drugs. 2017 Mar;77(3):247-264. doi: 10.1007/s40265-017-0694-4. PMID 28155046
- [Background] U.K. prospective diabetes study 16. Overview of 6 years' therapy of type II diabetes: a progressive disease. U.K. Prospective Diabetes Study Group. Diabetes. 1995 Nov;44(11):1249-58. PMID 7589820
- [Background] Levy J, Atkinson AB, Bell PM, McCance DR, Hadden DR. Beta-cell deterioration determines the onset and rate of progression of secondary dietary failure in type 2 diabetes mellitus: the 10-year follow-up of the Belfast Diet Study. Diabet Med. 1998 Apr;15(4):290-6. doi: 10.1002/(SICI)1096-9136(199804)15:43.0.CO;2-M. PMID 9585393
- [Background] Benford M, Milligan G, Pike J, Anderson P, Piercy J, Fermer S. Fixed-dose combination antidiabetic therapy: real-world factors associated with prescribing choices and relationship with patient satisfaction and compliance. Adv Ther. 2012 Jan;29(1):26-40. doi: 10.1007/s12325-011-0096-z. Epub 2012 Jan 12. PMID 22246944